CLINICAL TRIAL: NCT02047565
Title: A Two-part Study in Edoxaban-treated Healthy Subjects to Establish a Punch Biopsy Bleeding Model and to Evaluate the Effect of a 4-factor Prothrombin Complex Concentrate on Anticoagulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: DU176b-A-U158
Record Dates: First submitted 2013-12-02; First posted 2014-01-28 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2015-01

CONDITIONS: Bleeding
Keywords: punch biopsy
MeSH Terms: conditions — Hemorrhage | interventions — edoxaban; factor IX, factor VII, factor X, prothrombin drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part 1 - 60mg edoxaban (Experimental): Treatment A: single oral dose of 60 mg edoxaban (1 × 60 mg tablet)
  Interventions: Drug: 60mg edoxaban
- Part 1 - 180mg edoxaban (Experimental): Treatment B: single oral dose of 180 mg edoxaban (3 × 60 mg tablet)
  Interventions: Drug: 180mg edoxaban
- Part 2 - 60mg edoxaban and 50 IU/kg Beriplex P/N (Experimental): Dose cohort 1: 60 mg edoxaban + 50 IU/kg Beriplex P/N in 1 period and placebo (0.9% Sodium Chloride Injection, USP), in the other period
  Interventions: Drug: 60mg edoxaban; Drug: 50 IU/kg Beriplex P/N
- Part 2 - 60mg edoxaban and 20 IU/kg Beriplex P/N (Experimental): Dose cohort 2: 60 mg edoxaban + 25 IU/kg Beriplex P/N in 1 period and placebo (0.9% Sodium Chloride Injection, USP), in the other period
  Interventions: Drug: 60mg edoxaban; Drug: 25 IU/kg Beriplex P/N
- Part 2 - 60mg edoxaban and 10 IU/kg Beriplex P/N (Experimental): Dose cohort 3: 60 mg edoxaban + 10 IU/kg Beriplex P/N in 1 period and placebo (0.9% Sodium Chloride Injection, USP), in the other period
  Interventions: Drug: 60mg edoxaban; Drug: 10 IU/kg Beriplex P/N

INTERVENTIONS:
Drug: 60mg edoxaban
  Arms: Part 1 - 60mg edoxaban; Part 2 - 60mg edoxaban and 10 IU/kg Beriplex P/N; Part 2 - 60mg edoxaban and 20 IU/kg Beriplex P/N; Part 2 - 60mg edoxaban and 50 IU/kg Beriplex P/N
Drug: 180mg edoxaban
  Arms: Part 1 - 180mg edoxaban
Drug: 50 IU/kg Beriplex P/N
  Arms: Part 2 - 60mg edoxaban and 50 IU/kg Beriplex P/N
Drug: 25 IU/kg Beriplex P/N
  Arms: Part 2 - 60mg edoxaban and 20 IU/kg Beriplex P/N
Drug: 10 IU/kg Beriplex P/N
  Arms: Part 2 - 60mg edoxaban and 10 IU/kg Beriplex P/N

SUMMARY:
This Phase 1 study consists of 2 parts. Part 1 will be an open-label, randomized, 2 treatment, 2-way crossover study. Part 2 will be a double-blind (Sponsor unblinded), randomized, placebo controlled, sequential descending prothrombin complex concentrate dose, 2 sequence, 2 period crossover study. In both parts of the study, the assessor of BD and BV will remain blinded. In Part 2 of the study, both the subject and the clinic staff involved in study conduct will be blinded (with the exception of the pharmacist or nurse who prepares the blinded individual treatments from open-label supplies). The study programmer and statistician will also be blinded to treatment assignment. The Sponsor will remain unblinded for both parts of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects between 18 and 45 years of age, with a body mass index between 18 and 30 kg/m2, and weighing ≤ 110 kg.

Exclusion Criteria:

* Women of childbearing potential without proper contraceptive measures and women who are pregnant or breastfeeding. Women of childbearing potential who participate in the study must agree to use proper contraceptive measures from screening through 13 weeks after the last dose of study drug.
* Subjects with history of unexplained syncope. Subjects who have prior clearance of vasovagal events may be included.
* Subjects who have used any drugs or substances known to be strong inhibitors or strong inducers of cytochrome P450 (CYP) 3A4/5 enzymes or P-glycoprotein within 28 days prior to the first dosing.
* Subjects who have used any other nonprescription drugs (including herbal supplemental), except acetaminophen (up to 3 g/day) within 14 days prior to check-in.
* Subjects with history of major bleeding, major trauma, or major surgical procedure of any type within 6 months of dosing.
* Subjects with history of peptic ulcer, gastrointestinal bleeding (including hematemesis, melena, and rectal bleeding), or bleeding from hemorrhoids.
* Subjects with history of minor bleeding episodes such as epistaxis, rectal bleeding (spots of blood on toilet paper), and gingival bleeding within 3 months before the first dose.
* Subjects who have any family history, suspected or documented, of coagulopathy.
* Subjects who have participated in a previous edoxaban study within 6 months prior to the first dose.
* Subjects who used anticoagulants (eg, warfarin, low molecular weight heparin), antiplatelet agents (eg, clopidogrel), non-steroidal anti-inflammatory drugs, and/or acetylsalicylic acid 30 days prior to punch biopsy or who expect to use these during the study.
* Subjects with hemoglobin levels below 12 g/dL (men) or 11 g/dL (women) at screening.
* Subjects with creatinine clearance ≤ 80 mL/min (based on the Cockcroft-Gault equation).
* Subjects who are considered inappropriate for the punch biopsy procedure based on inability to visualize surface blood vessels, and history or likelihood of forming keloid scars.
* Subjects with known heparin-induced thrombocytopenia.
* Subjects who have a platelet count, PT, or INR outside of the normal range at baseline.
* Subjects with history or current evidence of clinically significant cardiac, hepatic, renal, pulmonary, endocrine, neurologic, infectious, gastrointestinal, hematologic, or oncologic disease as determined by screening history, physical examination, laboratory test results, or 12-lead electrocardiogram (ECG).

In addition, for Part 2:

* Subjects who are deficient in Factor V Leiden mutation.
* Subjects who are deficient in protein S, protein C, antithrombin, or factor II, or have prothrombin 20210A mutation.
* Subjects with known anaphylactic or severe systemic reactions to Beriplex P/N or any components in Beriplex P/N including heparin; FII, FVII, FIX, and FX; proteins C and S; antithrombin III; and human albumin.
* Subjects with current or history of disseminated intravascular coagulation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2013-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Bleeding duration 60mg edoxaban | Day 1
  To assess the variability and effect size of bleeding duration (BD) following punch biopsy in healthy subjects administered 60 mg edoxaban
Bleeding volume 60mg edoxaban | Day 1
  To assess the variability and effect size of bleeding volume (BV) following punch biopsy in healthy subjects administered 60 mg edoxaban
Bleeding duration 180mg edoxaban | Day 1
  To assess the variability and effect size of bleeding duration (BD) following punch biopsy in healthy subjects administered 180 mg edoxaban
Bleeding volume 180mg edoxaban | Day 1
  To assess the variability and effect size of bleeding volume (BV) following punch biopsy in healthy subjects administered 180 mg edoxaban

SECONDARY OUTCOMES:
Prothrombin Time | Day 1
  To evaluate the reversal of the effect of 60 mg edoxaban on Prothrombin Time (PT), International Normalized Ratio (INR), Activated Partial Thromboplastin Time (aPTT), and Thrombin Generation Assay (TGA) parameters by Beriplex P/N
International Normalized Ratio | Day 1
  To evaluate the reversal of the effect of 60 mg edoxaban on Prothrombin Time (PT), International Normalized Ratio (INR), Activated Partial Thromboplastin Time (aPTT), and Thrombin Generation Assay (TGA) parameters by Beriplex P/N
Activated Partial Thromboplastin Time | Day 1
  To evaluate the reversal of the effect of 60 mg edoxaban on Prothrombin Time (PT), International Normalized Ratio (INR), Activated Partial Thromboplastin Time (aPTT), and Thrombin Generation Assay (TGA) parameters by Beriplex P/N
Thrombin Generation Assay | Day 1
  To evaluate the reversal of the effect of 60 mg edoxaban on Prothrombin Time (PT), International Normalized Ratio (INR), Activated Partial Thromboplastin Time (aPTT), and Thrombin Generation Assay (TGA) parameters by Beriplex P/N
procoagulant markers D dimer | Day 1
  To evaluate the effects of Beriplex P/N following 60 mg edoxaban on the procoagulant markers D dimer and prothrombin fragment F1 + 2 (F1 + 2)
prothrombin fragment F1 + 2 | Day 1
  To evaluate the effects of Beriplex P/N following 60 mg edoxaban on the procoagulant markers D dimer and prothrombin fragment F1 + 2 (F1 + 2)
coagulation factor concentrations | Day 1
  To evaluate the effects of Beriplex P/N following 60 mg edoxaban on coagulation factor concentrations
cmax of edoxaban and its active metabolite, D21-2393 | Day 1
  To evaluate single dose pharmacokinetics (PK) of edoxaban and its active metabolite, D21-2393
tmax of edoxaban and its active metabolite, D21-2393 | Day 1
  To evaluate single dose pharmacokinetics (PK) of edoxaban and its active metabolite, D21-2393
AUC 0-24 of edoxaban and its active metabolite, D21-2393 | Day 1
  To evaluate single dose pharmacokinetics (PK) of edoxaban and its active metabolite, D21-2393

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Zahir H, Brown KS, Vandell AG, Desai M, Maa JF, Dishy V, Lomeli B, Feussner A, Feng W, He L, Grosso MA, Lanz HJ, Antman EM. Edoxaban effects on bleeding following punch biopsy and reversal by a 4-factor prothrombin complex concentrate. Circulation. 2015 Jan 6;131(1):82-90. doi: 10.1161/CIRCULATIONAHA.114.013445. Epub 2014 Nov 17. PMID 25403645